CLINICAL TRIAL: NCT06498167
Title: Active Pharmacovigilance Study of the Medicine Rinvoq™ (Upadacitinib)
Acronym: LOOK-UP
Status: Recruiting | Type: Observational
Sponsor: Universidade do Porto (Other)
Collaborators: INFARMED - Autoridade Nacional do Medicamento e Produtos de Saúde, I.P. (Unknown); Unidade de Farmacovigilância do Porto (Unknown); Unidade Local de Saúde São João (Other Government); Unidade Local de Saúde de Santo António, E.P.E. (Unknown); Unidade Local de Saude de Gaia e Espinho EPE (Other); RISE Health (Unknown)
Responsible Party: Sponsor
Other Study IDs: LookUp; EUPAS1000000227 (Other: European Medicines Agency)
Record Dates: First submitted 2024-07-04; First posted 2024-07-12 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Inflammatory Disease; Drug Side Effect; Drug Use; Adverse Drug Event; Adverse Drug Reaction; Safety Issues
Keywords: Upadacitinib; Rinvoq; Rheumatoid arthritis; Psoriatic arthritis; Axial spondyloarthritis; Atopic dermatitis; Ulcerative colitis; Crohn's disease; Pharmacovigilance risk; Drug safety monitoring; Patient Safety
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Arthritis, Rheumatoid; Arthritis, Psoriatic; Axial Spondyloarthritis; Dermatitis, Atopic; Colitis, Ulcerative; Crohn Disease | interventions — upadacitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Upadatacinib Arm: Patients exposed to upadacitinib (Rinvoq™)
  Interventions: Drug: Upadacitinib

INTERVENTIONS:
Drug: Upadacitinib — Exposure to upadacitinib (Rinvoq™) in its different formulations approved by the Portuguese regulatory authority (15, 30, or 45mg extended-release tablets).
  Other Names: Rinvoq; ATC 200000041628

SUMMARY:
The LOOK-UP is an investigator-initiated clinical study with the aim of monitoring the post-marketing safety of the medicine Rinvoq™ (upadacitinib), which is indicated for the treatment of rheumatoid arthritis, psoriatic arthritis, axial spondyloarthritis, atopic dermatitis, ulcerative colitis, and Crohn's disease. The Marketing Authorisation Holder is AbbVie Deutschland GmbH & Co. KG.

DETAILED DESCRIPTION:
The LOOK-UP study is an investigator-initiated clinical study conducted by INFARMED, the Portuguese Authority of Medicines and Health Products, I.P., and coordinated by the Porto Pharmacovigilance Centre at the Faculty of Medicine, University of Porto. The study aims to monitor the post-marketing safety of Rinvoq™ (upadacitinib), a medicine indicated for the treatment of rheumatoid arthritis, psoriatic arthritis, axial spondyloarthritis, atopic dermatitis, ulcerative colitis, and Crohn's disease. Rinvoq™, a selective and reversible Janus Kinase (JAK) 1 inhibitor, has been under additional monitoring by the European Medicines Agency (EMA) since its approval in December 2019, necessitating active safety surveillance in real-world settings.

The primary objective of the LOOK-UP study is to quantify the incidence of adverse events in patients prescribed Rinvoq™, with a focus on serious adverse events such as malignant neoplasms, non-melanoma skin cancer, major adverse cardiovascular events, venous thromboembolism, serious and opportunistic infections, gastrointestinal perforations, liver injuries, bone fractures, and all-cause mortality. Secondary objectives include describing the incidence of adverse events among specific subgroups, such as very elderly patients, patients with moderate hepatic impairment, and patients with severe renal impairment. Additionally, the study aims to characterize patient-reported adverse events using MedDRA terms. An exploratory objective is to evaluate adherence to risk minimization measures recommended by the Pharmacovigilance Risk Assessment Committee (PRAC) for the safe use of Rinvoq™.

The study is designed as a Phase 4 post-authorization safety study (PASS), utilizing an observational cohort approach that is both multicentric and ambispective. This design includes prospective and retrospective monitoring of patients, ensuring comprehensive safety analysis. The study will be conducted exclusively in hospital settings within the Porto district, reflecting the prescription and usage constraints of Rinvoq™.

ELIGIBILITY:
Inclusion Criteria:

* Prescription of Rinvoq™ from January 1, 2024;
* 18 years of age or older at the time of recruitment; and
* Expressed consent to participate in the study.

Exclusion Criteria:

* They have any degree of cognitive impairment that prevents them from responding to a questionnaire administered by telephone;
* They are participating in a phase I, II, or III clinical trial;
* They have a life expectancy of less than 1 month; or
* They do not have a valid telephone contact.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients exposed to upadacitinib (Rinvoq™).
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | For the prospective cohort, the follow-up includes contacts at baseline (t=0), 2 weeks (t=1), 1 month (t=2), 2 months (t=3), and 3 months (t=4) after starting treatment.
  Incidence of adverse events occurring during the established follow-up period, coded according to MedDRA terminology.
  The outcome will be assessed through an ad-hoc questionnaire. The occurrence of adverse events will be queried in an open-ended, non-directed manner. Patients will be encouraged to report any undesired events they experience during the treatment, without being limited to predefined specific adverse events.

SECONDARY OUTCOMES:
Rate of non-compliance with PRAC recommendations | This outcome will be assessed at any time during the three-month monitoring period of each patient.
  Rate at which patients identified with risk factors are prescribed Rinvoq™ despite the availability of viable therapeutic alternatives. Patients considered to have risk factors include: (i) individuals aged 65 or older; (ii) current smokers or those with a long history of smoking; (iii) individuals at high risk of serious cardiovascular problems, such as heart attacks or strokes, or those more likely to develop cancer.
  The outcome will be assessed through direct contact with clinical specialists (prescribers) to confirm the availability of therapeutic alternatives. A case is non-compliant if a patient with risk factors is prescribed Rinvoq™ despite an available alternative.

CONTACTS AND LOCATIONS:
Overall Officials: Inês Ribeiro Vaz, PharmD, MPH, PhD, Principal Investigator — Universidade do Porto
Locations (3):
- Portugal (3):
  - Unidade Local de Saúde de Santo António, E.P.E., Porto
  - Unidade Local de Saúde de São João, E.P.E., Porto
  - Unidade Local de Saúde de Gaia/Espinho, E.P.E., Porto